CLINICAL TRIAL: NCT06307951
Title: Exploration of Infant and Young Child Feeding Practices and Their Determinants Among Women Living in Urban Areas and Slums in Pune and Rural Areas Around Pune, India
Brief Title: Exploration of Infant and Young Child Feeding Practices and Their Determinants
Status: Completed | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: JCDC/BHR/24/012
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to assess infant and young child-feeding practices among women living in urban areas and slums in Pune and rural areas around Pune, India, and to investigate the reasons for the adopted infant and young child-feeding practices in Slum-dwelling women aged 18 to 49 years who have an infant/s less than 24 months of age.

The main question it aims to answer are:

* Are infant and young child-feeding practices among women living in urban areas and slums appropriate?
* What the reasons for the adopted infant and young child-feeding practices in Slum-dwelling women Participants will be measured for their height and weight, interviewed for Socio-demographic characteristics, birth history of the infant, infant feeding indicators and will be involved in focused group discussions and in-depth interviews to gain understanding into their adopted appropriate and inappropriate feeding practices.

DETAILED DESCRIPTION:
Study Design: Cross-sectional, Observational Study Duration: 2 years Population Characteristics: Slum-dwelling women aged 18 to 49 years who have an infant/s less than 24 months of age Study Site / Subject Recruitment: Subjects will be recruited at the family planning department of urban health care centres and Paediatric OPDs in tertiary care hospitals in the Pune city and rural health care centres around Pune city where they take their children for vaccination

ELIGIBILITY:
Inclusion Criteria:

* A woman will be recruited in the study if she

  1. is willing and able to give informed consent
  2. is aged between 18 to 49 years
  3. has an infant or infants less than 2 years of age

Exclusion Criteria:

1. She is unwilling to consent to participate in the study
2. Her infant has any congenital conditions, chronic disorder or has a disorder resulting in difficulty in feeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Slum-dwelling women aged 18 to 49 years who have an infant/s less than 24 months of age
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Infant and young child-feeding practices among women living in urban areas and slums in Pune and rural areas around Pune, India will have been assessed | 2 years
  Infant and young child-feeding practices among women living in urban areas and slums in Pune and rural areas around Pune, India will have been assessed

SECONDARY OUTCOMES:
Reasons for the adopted infant and young child-feeding practices will have been investigated | 2 years
  Reasons for the adopted infant and young child-feeding practices will have been investigated

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Khadilkar, M.D., Principal Investigator — Hirabai Cowasji Jehangir Medical Research Institute
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No